CLINICAL TRIAL: NCT01050348
Title: A Double Blinded Randomized Placebo Controlled Study: To Investigate the Role of Upstream High Dose Statin Treatment in Patients With ST Segment Elevation Myocardial Infarction
Brief Title: To Investigate the Role of Upstream High Dose Statin in STEMI
Acronym: IMPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Western Pennsylvania Hospital (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-004 / WPCI 2009-08
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin calcium (Active Comparator): Patients will receive study medication upon admission to hospital prior to percutaneous intervention of the culprit artery
  Interventions: Drug: Atorvastatin calcium
- Sugar Pill (Placebo Comparator): Patients will receive study medication upon admission to hospital prior to percutaneous intervention of the culprit artery
  Interventions: Drug: Inactive Placebo

INTERVENTIONS:
Drug: Atorvastatin calcium — Eligible patients will receive 80mgs of atorvastatin orally upon admission to hospital prior to percutaneous intervention of the affected artery. Dose of post-procedural statin will be at the discretion of the cardiologist.
  Other Names: Lipitor
  Arms: Atorvastatin calcium
Drug: Inactive Placebo — Eligible patients will receive a placebo orally upon admission to hospital prior to percutaneous intervention of the affected artery.
  Other Names: Placebo, Sugar Pill
  Arms: Sugar Pill

SUMMARY:
This is a double-blinded randomized placebo controlled trial investigating the role of upstream 80mg Atorvastastin-calcium in patients undergoing percutaneous intervention for acute STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient of 25 to 90 years of age admitted or transferred to Western Pennsylvania Hospital or Allegheny General Hospital with a diagnosis of STEMI undergoing emergent percutaneous intervention (PCI) to the culprit coronary artery. STEMI is defined as greater than 1mm ST segment elevation on electrocardiogram.
2. Elevated cardiac biomarkers (troponin-T > 0.03ng/ml, CKMB>5ng/mL, or ck>170 U/l).

Exclusion Criteria:

1. Known history of liver disease defined as cirrhosis, alcoholic liver disease, Non alcoholic steatohepatitis, hepatitis or any causes of liver failure.
2. Renal failure with creatinine >3mg/dL
3. Known history of liver or muscle disease such as rheumatologic myopathies, history of myositis, hepatitis, and hepatic cancer.
4. Cardiovascular arrest and shock.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) defined as cardiovascular death, MI, or target revascularization 30 days post percutaneous intervention. | 15 and 30 days post revascularization

SECONDARY OUTCOMES:
Any increase in mean peak values of CK-MB, troponin I and myoglobin greater than twice the upper limit after intervention. | 15 and 30 days post revascularization
Any occurrence of major adverse cardiac events defined as death, MI, congestive heart failure, cardiogenic shock or need for unplanned revascularization within 24 hours after procedure or need for emergent CABG. | 15 and 30 days post revascularization
Symptomatic side effects of current statin medication as described by adverse effects on consent form. | Immediately post revascularization to 30 days.
Modified Coronary Revascularization Outcome Questionnaire (CROQ-PTCA) | 15 and 30 days post revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Venkatraman Srinivasan, MD, Principal Investigator — West Penn Allegheny Health System
Locations (2):
- United States (2):
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania